CLINICAL TRIAL: NCT03366064
Title: Phase I Trial of Haploidentical Natural Killer (NK) Cells in Combination With Pemetrexed in Patients With Stage IV Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Haploidentical NK Cells After Pemetrexed in Patients With Stage IV Non-Small Cell Lung Cancer (NSCLC)
Acronym: Medi-NK
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Collaborators: Korea Research Institute of Bioscience & Biotechnology (Other Government)
Responsible Party: Principal Investigator, Kyoo-Hyung Lee, Professor, Hematology, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-0607
Record Dates: First submitted 2017-12-04; First posted 2017-12-08 (Actual); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Non-small cell lung cancer; Natural killer cells; HLA-haploidentical family donor
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pemetrexed and donor NK cell infusion (Experimental): Eligible patients with stage 4 non-small cell lung cancer receive NK cells derived from HLA-haploidentical family donors. One week prior to NK cell infusion, patients receive pemetrexed (500 mg/m2) intravenous infusion
  Interventions: Biological: Pemetrexed and donor-derived NK cell infusion

INTERVENTIONS:
Biological: Pemetrexed and donor-derived NK cell infusion — Patients are administered with donor-derived NK cells one week after pemetrexed infusion

SUMMARY:
This phase 1 trial investigate safety and maximum tolerated dose of natural killer (NK) cells derived from haploidentical family donors in patients with non-small cell lung cancer

DETAILED DESCRIPTION:
Eligible patients receive pemetrexed 500 mg/m2 intravenously (Day 1). On Day 8, patients receive donor-derived NK cells via a central venous catheter.

The NK cell dose is as follows;

Level 1: 1.25 X 109 cells Level 2: 2.50 X 109 cells Level 3: 5.00 X 109 cells

Three patients each will be treated on each dose level.

Two weeks prior to donor NK cell administration to patients, HLA-haploidentical family member of the patients undergo leukapheresis after G-CSF injections to collect hematopoietic stem cells.

These donor cells are then taken to the laboratory, where they were differentiated into NK cells ex vivo over approximately over 2-week period.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed non-small cell lung cancer stage 4 (by AJCC 7th)
* Age, 20 years of age or older
* ECOG performance status, 0-2
* Life expectancy ≥3 months
* Patients should have at least one measurable lesion according to RECIST Criteria v1.1
* Failure after primary systemic treatment with a regimen including platinum-containing agent (primary systemic treatment may be adjuvant chemotherapy or chemo-radiotherapy, given within 12 months)
* Adequate bone marrow function (Hb ≥9 g/dL; ANC ≥1,500/uL; and platelet count ≥75,000/uL)
* Adequate renal function (serum creatinine <1 x ULN or CLcr ≥45 mL/min by Cockroft and Gault formula
* Adequate liver function (total bilirubin <1.5 x ULN; AST and ALT <3 x ULN; and ALP <3 x ULN, unless there is bone metastases without evidence of liver disease)
* Patients should have a suitable HLA-haploidentical family member who is willing to donate hematopoietic stem cells
* Patients should sign informed consent voluntarily

Exclusion Criteria:

* Patients who received anti-cancer chemotherapeutic or biological agents within 3 weeks. Patients who received anti-cancer treatment and did not recover from toxicities to grades 0-1 by NCI CTC AE ver 4.0 are not eligible as well.
* Patients with contraindication for any medication planned to be administered in the study
* Patients with significant fluid accumulation in third space (for example, pleural or pericardial effusion) that can not be controlled by drainage
* Active infectious process
* Inability to discontinue aspirin over 1.3 g daily or other NSAIDs. Patients cannot take aspirin or NSAIDs within 5 days of pemetrexed administration
* Major surgery within 4 weeks of study participation
* Palliative radiation therapy within 1 week of study participation
* Acute myocardial infarction within 6 months of study participation. History of uncontrolled arrhythmia, symptomatic angina, or symptomatic heart failure
* Past or current history of CNS metastasis (with exception of those patients who completed treatment of CNS metastasis and not received steroid treatment or whole brain radiotherapy within 2 weeks of screening visit or not received gamma knife treatment within 1 week of screening visit)
* History of malignancy (other than skin basal cell carcinoma, carcinoma in situ of uterine cervix, or thyroid cancer) within 5 years
* Pregnant or lactating women. Child-bearing women who are not willing to avoid pregnancy by contraceptives
* Man not agreeing to contraceptive measures such as condom or abstinence (It is recommended that contraceptive measures be used until 6 months after pemetrexed treatment)
* Other serious illness or medical condition

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2017-11-09 (Actual); Primary Completion 2018-09-03 (Actual); Study Completion 2019-06-15 (Actual)

PRIMARY OUTCOMES:
maximum tolerated dose of donor NK cells | 6 weeks
  determine the dose of NK cells that can be given within dose-limiting toxicities

CONTACTS AND LOCATIONS:
Overall Officials: Kyoo-Hyung Lee, MD, Principal Investigator — University of Ulsan, Asan Medical Center
Locations (1):
- Asan Medical Center - University of Ulsan College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yoon SR, Lee YS, Yang SH, Ahn KH, Lee JH, Lee JH, Kim DY, Kang YA, Jeon M, Seol M, Ryu SG, Chung JW, Choi I, Lee KH. Generation of donor natural killer cells from CD34(+) progenitor cells and subsequent infusion after HLA-mismatched allogeneic hematopoietic cell transplantation: a feasibility study. Bone Marrow Transplant. 2010 Jun;45(6):1038-46. doi: 10.1038/bmt.2009.304. Epub 2009 Nov 2. PMID 19881555
- [Background] Lee KH, Lee JH, Lee JH, Kim DY, Park HS, Choi EJ, Ko SH, Seol M, Lee YS, Kang YA, Jeon M, Baek S, Kang YL, Kim SH, Yun SC, Kim H, Jo JC, Choi Y, Joo YD, Lim SN. Reduced-Intensity Conditioning with Busulfan, Fludarabine, and Antithymocyte Globulin for Hematopoietic Cell Transplantation from Unrelated or Haploidentical Family Donors in Patients with Acute Myeloid Leukemia in Remission. Biol Blood Marrow Transplant. 2017 Sep;23(9):1555-1566. doi: 10.1016/j.bbmt.2017.05.025. Epub 2017 May 25. PMID 28552421
- [Background] Choi I, Yoon SR, Park SY, Kim H, Jung SJ, Jang YJ, Kang M, Yeom YI, Lee JL, Kim DY, Lee YS, Kang YA, Jeon M, Seol M, Lee JH, Lee JH, Kim HJ, Yun SC, Lee KH. Donor-derived natural killer cells infused after human leukocyte antigen-haploidentical hematopoietic cell transplantation: a dose-escalation study. Biol Blood Marrow Transplant. 2014 May;20(5):696-704. doi: 10.1016/j.bbmt.2014.01.031. Epub 2014 Feb 11. PMID 24525278
- [Background] Lee KH, Lee JH, Lee JH, Kim DY, Seol M, Lee YS, Kang YA, Jeon M, Hwang HJ, Jung AR, Kim SH, Yun SC, Shin HJ. Reduced-intensity conditioning therapy with busulfan, fludarabine, and antithymocyte globulin for HLA-haploidentical hematopoietic cell transplantation in acute leukemia and myelodysplastic syndrome. Blood. 2011 Sep 1;118(9):2609-17. doi: 10.1182/blood-2011-02-339838. Epub 2011 Jun 28. PMID 21715313
- [Background] Choi I, Yoon SR, Park SY, Kim H, Jung SJ, Kang YL, Lee JH, Lee JH, Kim DY, Lee JL, Park HS, Choi EJ, Lee YS, Kang YA, Jeon M, Seol M, Baek S, Yun SC, Kim HJ, Lee KH. Donor-Derived Natural Killer Cell Infusion after Human Leukocyte Antigen-Haploidentical Hematopoietic Cell Transplantation in Patients with Refractory Acute Leukemia. Biol Blood Marrow Transplant. 2016 Nov;22(11):2065-2076. doi: 10.1016/j.bbmt.2016.08.008. Epub 2016 Aug 12. PMID 27530969